CLINICAL TRIAL: NCT02451982
Title: A Platform Study of Combination Immunotherapy for the Neoadjuvant and Adjuvant Treatment of Patients With Surgically Resectable Adenocarcinoma of the Pancreas
Brief Title: Platform Study of Neoadjuvant and Adjuvant Immunotherapy for Patients With Resectable Adenocarcinoma of the Pancreas
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1568; IRB00050517 (Other: JHMIRB); R01CA197296 (NIH)
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cyclophosphamide; Nivolumab; urelumab; HuMax-IL8

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A: CY/GVAX alone (Experimental): Patients receive low-dose cyclophosphamide IV on day 0 and GVAX pancreatic cancer vaccine ID on day 1. Patients undergo pancreaticoduodenectomy on day 15. Approximately 6-10 weeks after surgery, patients receive low-dose cyclophosphamide IV on day 0 and the vaccine on day 1. Beginning approximately 1 month after vaccination, patients receive standard adjuvant chemoradiotherapy. Beginning approximately 4-8 weeks after the completion of chemoradiotherapy, patients receive low-dose cyclophosphamide IV on day 0 and the vaccine on day 1. Treatment with cyclophosphamide and the vaccine repeats every 28 days for 4 courses. Patients will then enter the extended treatment phase where they will receive cyclophosphamide on day 0, and GVAX on day 1 every 12 weeks for another 2 treatments.
  Interventions: Drug: Cyclophosphamide; Biological: GVAX pancreatic cancer
- Arm B: CY/GVAX with nivolumab (Experimental): Patients receive low-dose cyclophosphamide and nivolumab IV on day 0 and GVAX pancreatic cancer vaccine ID on day 1. Patients undergo pancreaticoduodenectomy on day 15. Approximately 6-10 weeks after surgery, patients receive low-dose cyclophosphamide and nivolumab IV on day 0 and the vaccine on day 1. Beginning approximately 1 month after vaccination, patients receive standard adjuvant chemoradiotherapy. Beginning approximately 4-8 weeks after the completion of chemoradiotherapy, patients receive low-dose cyclophosphamide and nivolumab IV on day 0 and the vaccine on day 1. Treatment with cyclophosphamide, nivolumab, and the vaccine repeats every 28 days for 4 courses. Patients will then enter the extended treatment phase where they will receive nivolumab every 4 weeks for another 6 treatments as well as cyclophosphamide on day 0, and GVAX on day 1 every 12 weeks for another 2 treatments.
  Interventions: Drug: Cyclophosphamide; Biological: GVAX pancreatic cancer; Drug: Nivolumab
- Arm C: CY/GVAX with nivolumab and urelumab (Experimental): Patients receive low-dose cyclophosphamide, nivolumab, and urelumab on day 0 and GVAX pancreatic cancer vaccine on day 1. Patients undergo pancreaticoduodenectomy on day 15. Approximately 6-10 weeks after surgery, patients receive low-dose cyclophosphamide, nivolumab, and urelumab on day 0 and the vaccine on day 1. Beginning approximately 28 days after vaccination, patients receive standard adjuvant chemoradiotherapy. Beginning approximately 4-8 weeks after the completion of chemoradiotherapy, patients receive low-dose cyclophosphamide, nivolumab, and urelumab on day 0 and GVAX on day 1. Treatment with cyclophosphamide, nivolumab, urelumab, and the vaccine repeats every 28 days for 4 courses. Patients will then enter the extended treatment phase where they will receive nivolumab and urelumab every 4 weeks for another 6 treatments as well as cyclophosphamide on day 0, and GVAX on day 1 every 12 weeks for another 2 treatments.
  Interventions: Drug: Cyclophosphamide; Biological: GVAX pancreatic cancer; Drug: Nivolumab; Drug: Urelumab
- Arm D: BMS-986253 and Nivolumab (Experimental): Patients receive BMS-986253 and nivolumab on day 0 (Cycle 1), 15 days prior to surgery. 6-10 weeks after surgery, patients receive Cycle 2, with nivolumab on day 0 and BMS-986253 on days 0 and 14. Patients then receive standard adjuvant chemoradiotherapy. Approximately 4-8 weeks after the completion of chemoradiotherapy, patients receive 4 additional 28-day cycles of immunotherapy, with Nivolumab on Day 0 and BMS-986253 on Days 0 and 14. Patients will then enter the extended treatment phase where they will receive nivolumab alone every 4 weeks for another 6 treatments.
  Interventions: Drug: Nivolumab; Drug: BMS-986253

INTERVENTIONS:
Drug: Cyclophosphamide — 200 mg/m2 IV
  Other Names: Cytoxan, CY
  Arms: Arm A: CY/GVAX alone; Arm B: CY/GVAX with nivolumab; Arm C: CY/GVAX with nivolumab and urelumab
Biological: GVAX pancreatic cancer — 5x10^8 cells intradermal injection
  Other Names: GVAX, pancreatic tumor vaccine
  Arms: Arm A: CY/GVAX alone; Arm B: CY/GVAX with nivolumab; Arm C: CY/GVAX with nivolumab and urelumab
Drug: Nivolumab — 480 mg IV
  Other Names: OPDIVO; BMS-936558; anti-PD1
  Arms: Arm B: CY/GVAX with nivolumab; Arm C: CY/GVAX with nivolumab and urelumab; Arm D: BMS-986253 and Nivolumab
Drug: Urelumab — 8 mg IV
  Other Names: BMS-663513; anti-CD137 Agonist
  Arms: Arm C: CY/GVAX with nivolumab and urelumab
Drug: BMS-986253 — 2400 mg IV
  Other Names: anti-IL8 antibody; HuMax-IL8
  Arms: Arm D: BMS-986253 and Nivolumab

SUMMARY:
This platform trial will evaluate various immunotherapy combinations given in the neo-adjuvant and adjuvant setting in patients with surgically resectable pancreatic ductal adenocarcinoma.

DETAILED DESCRIPTION:
Immunotherapy is an innovative approach being developed for the treatment of pancreatic cancer, a lethal and relatively chemotherapy-resistant disease. However, the tumor and its environment have developed a number of ways in which they inhibit the function of the immune system preventing it from recognizing and killing the cancer. In addition, the investigators still do not understand how T cells, the cells in the immune system that have the potential to recognize cancer as different and kill cancer cells, traffic into the tumor to accomplish their task. The investigators are currently testing an immune system activating pancreatic cancer vaccine (known as GVAX) in combination with immune boosting doses of the chemotherapy agent, cyclophosphamide, as preoperative and postoperative treatments for pancreatic cancer. The investigators have discovered tertiary lymphoid aggregates, a unique lymph node-like structure formed within resected tumors from the patients who received the vaccine two weeks prior to the surgery. This discovery demonstrates that the immune system can get into the tumor and provides the investigators with the opportunity to better understand how these immune cells traffic into the tumor and function once they arrive. The investigators also found that the vaccine causes an increase in signals that would suppress the immune system's ability to fight off cancer cells, including signals involving PD-1. In this novel study, the investigators will test the effects of blocking PD-1 in combination with the vaccine in patients with pancreatic cancer. The investigators will specifically isolate these immune cells and evaluate at both the genetic and protein level, the types of signals expressed by these aggregates. The investigators will compare aggregates from patients with long term survival versus patients who succumb to their cancer early. In this way, the investigators will be able to determine how safe this novel treatment is, how effective it is at changing the immune system in pancreatic cancer, and how it impacts the health and survival of pancreatic cancer patients who undergo surgery to remove the cancer.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or clinically-suspected adenocarcinoma of the head, neck, or uncinate process of the pancreas
* Tumor must be surgically resectable
* ECOG Performance Status of 0 to 1
* Adequate organ function as defined by study-specified laboratory tests
* Must agree to use acceptable form of birth control

Exclusion Criteria:

* Received any type of anti-cancer treatment or immunotherapy for pancreas cancer
* History of autoimmune disease (Graves or Hashimoto's disease, vitiligo, and type I diabetes are allowed)
* Systemically steroid use within 14 days
* Evidence of active infection
* Pregnant or lactating
* Diagnosed with another cancer or myeloproliferative disorder (some exceptions)
* History of severe hypersensitivity reaction to any monoclonal antibody or known component of the study drugs
* Known history of infection with HIV, hepatitis B, or hepatitis C
* Oxygen saturation of <92% on room air by pulse oximetry
* On home oxygen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2016-03-28 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
IL17A expression | 4 years
  median IL17A expression in lymphoid aggregates from resected tumor (Arms A and B only)
Intratumoral CD8+CD137+cells | 4 years
  Fold change of intratumoral CD8+CD137+cells before and after neoadjuvant therapy (Arms B and C only)
Intratumoral granzyme B+PD-1+CD137+ cells | 4 years
  Percent change of intratumoral granzyme B+PD-1+CD137+ cells in surgical (post-treatment) tissue compared to baseline (pre-treatment) biopsy (Arm D only)
Pathologic Response | 4 years
  Percent of patients with a response grade of 0-2 (0=complete response 1=marked response, 2=moderate response) at time of surgery

SECONDARY OUTCOMES:
Drug-Related Adverse Events | 4 years
  Number of participants experiencing study drug-related toxicities
Overall Survival | 4 years
  Overall Survival is defined as the time from surgery to death from any cause
Disease Free Survival | 4 years
  Disease Free Survival is defined as the time from surgery until evidence of disease recurrence or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Ana De Jesus-Acosta, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Heumann T, Judkins C, Li K, Lim SJ, Hoare J, Parkinson R, Cao H, Zhang T, Gai J, Celiker B, Zhu Q, McPhaul T, Durham J, Purtell K, Klein R, Laheru D, De Jesus-Acosta A, Le DT, Narang A, Anders R, Burkhart R, Burns W, Soares K, Wolfgang C, Thompson E, Jaffee E, Wang H, He J, Zheng L. A platform trial of neoadjuvant and adjuvant antitumor vaccination alone or in combination with PD-1 antagonist and CD137 agonist antibodies in patients with resectable pancreatic adenocarcinoma. Nat Commun. 2023 Jun 20;14(1):3650. doi: 10.1038/s41467-023-39196-9. PMID 37339979